CLINICAL TRIAL: NCT00335907
Title: Protocol-driven Hemodynamic Support for Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Jonathan Sevransky, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-23 NIGMS 2005
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Shock, Septic; Severe Sepsis; Sepsis
Keywords: Clinical trial; Controlled clinical trial; Shock, Septic
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Fluid Therapy

INTERVENTIONS:
Procedure: Fluid and Vasopressor Protocol — A Physician Ordered, Nurse Administered Fluid and Vasopressor Protocol

SUMMARY:
This research is being done to see if a protocol (a set of orders that determine how much and how quickly a drug/fluid is given) for fluid and drugs used to increase blood pressure (vasopressors) will work better then general clinical practices to improve outcomes in patients with septic shock.

DETAILED DESCRIPTION:
Septic shock is low blood pressure caused by an infection. Sepsis is the most common cause of death in non-cardiac intensive care units, and septic shock is the most severe form of sepsis. Treatment for septic shock includes giving antibiotics, intravenous fluids, and medications to raise the blood pressure (vasopressors).

We would like to see if a protocol-driven management strategy for septic shock can shorten time on vasopressors and limit the number of side effects. We have constructed a protocol that will allow the nurse at the bedside, in conjunction with the physician's orders, to adjust the amount of fluids and medications that raise the blood pressure (vasopressors).

ELIGIBILITY:
Inclusion Criteria:

* ACCP/SCCM sepsis criteria
* Need for institution of vasopressors after adequate volume resuscitation

Exclusion Criteria:

* Age< 18
* On vasopressors for > 24 hours prior to ICU admission
* Other cause for shock ( cardiac tamponade, massive pulmonary embolus, cardiogenic shock)
* Physicians and family not committed to aggressive medical therapy ( a patient will not be excluded if he/she would receive all care except for attempts at resuscitation from cardiac arrest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-06 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Length of vasopressor treatment | within 90 days

SECONDARY OUTCOMES:
Total number of vials vasopressors administered | Within 90 days
Time on more than single vasopressor | Within 90 days
Volume of intravenous fluids administered in first 7 days | 7 days
Number of organ failures | Within 90 days
ICU mortality rates | Within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Sevransky, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States